CLINICAL TRIAL: NCT00236769
Title: An Open-label Study to Evaluate Contraceptive Efficacy and Safety of the Transdermal Contraceptive System of 17deacetyl-norgestimate and Ethinyl Estradiol.
Brief Title: A Study of Efficacy and Safety With the Transdermal Contraceptive System.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR005500
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2010-11-17 (Estimated); Status verified 2010-11

CONDITIONS: Contraception; Female Contraception
Keywords: contraception; transdermal contraception; hormonal, steroidal contraception; ethinyl estradiol; progesterone
MeSH Terms: interventions — norelgestromin; Ethinyl Estradiol

INTERVENTIONS:
Drug: norelgestromin + ethinyl estradiol

SUMMARY:
The purpose of the study is to evaluate the contraceptive efficacy, safety, cycle control, and compliance with the transdermal contraceptive system.

DETAILED DESCRIPTION:
This is an open-label, multicenter, global study to evaluate the contraceptive efficacy, cycle control, safety, compliance and subject satisfaction of the transdermal contraceptive system. Sixteen hundred healthy women will wear the contraceptive patch for either 6 or 13 cycles. The first 530 subjects will wear the patch for 13 cycles, and all subsequent subjects will wear the patch for 6 cycles. At admission Visit 1, study drug (plus 3 reserve patches) and diary cards are dispensed for Cycle 1; first patch application will be on the first day of menses. Study drug and diary cards are dispensed on day 28 of Cycle 1 (Visit 2) for Cycles 2 and 3, on day 28 of Cycle 3 (Visit 3) for Cycles 4 to 6, on day 28 of Cycle 6 (Visit 4) for Cycles 7 to 9, and on day 28 of Cycle 9 (Visit 5) for Cycles10 to13. At each of these visits, diary cards and empty medication packages are collected. Final study visits are on day 28 of Cycles 6 and 13. Diary card information is used to record compliance and bleeding information (to assess cycle control). Contraceptive efficacy is assessed by means of the Pearl Index and life table analysis (gross cumulative probability of pregnancy). Safety evaluations are based on adverse events, which are collected throughout the study, and changes in gynecologic examinations, vital signs, and laboratory results from admission to final visit. Each transdermal contraceptive patch, containing 6 mg NGM and 0.75 mg EE, and delivering 250 ug 17-dNGM and 25 ug EE over 24 hours for 7 days, is worn for 1 week and replaced for 3 consecutive weeks. The fourth week is patch-free. The patch can be worn on: upper arm or torso, buttock, or abdomen.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women with regular menstrual cycles
* sexually active and at risk of pregnancy
* nonpregnant
* acceptable body mass index (BMI)
* last term pregnancy at least 42 days prior, nonlactating, with 1 normal menstrual cycle since
* sitting BP<140mmHg/<90mmHg
* 1 normal menstrual cycle since removal of IUD or norplant
* agreement to use study drug for contraception for up to 13 cycles, except when backup contraception is required for disease protection or patch detachment
* agree not to use other systemic steroid medication

Exclusion Criteria:

* Presence, history, hereditary predisposition or risk of deep vein thrombophlebitis or thromboembolic disorders
* cerebral vascular or coronary artery disease, hypertension, or severe migraines
* liver tumor resulting from estrogen-containing products
* diabetes mellitus
* cholestatic jaundice, liver or renal disease
* abnormal PAP smear
* thyroid disorder
* dermal hypersensitivity
* carcinoma of breast, endometrium or other estrogen-dependent neoplasia
* substance abuse
* received experimental drug within prior 30 days
* smoking women over 35 years of age.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1751 (Actual)
Dates: Start 1997-11; Study Completion 1999-10 (Actual)

PRIMARY OUTCOMES:
Contraceptive efficacy is assessed with the Pearl Index and life table analysis (gross cumulative probability of pregnancy). Safety is evaluated throughout the study.

SECONDARY OUTCOMES:
Cycle control and compliance are assessed with diary cards containing bleeding information and dosing information.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Smallwood GH, Meador ML, Lenihan JP, Shangold GA, Fisher AC, Creasy GW; ORTHO EVRA/EVRA 002 Study Group. Efficacy and safety of a transdermal contraceptive system. Obstet Gynecol. 2001 Nov;98(5 Pt 1):799-805. doi: 10.1016/s0029-7844(01)01534-4. PMID 11704172
- [Result] Zieman M, Guillebaud J, Weisberg E, Shangold GA, Fisher AC, Creasy GW. Contraceptive efficacy and cycle control with the Ortho Evra/Evra transdermal system: the analysis of pooled data. Fertil Steril. 2002 Feb;77(2 Suppl 2):S13-8. doi: 10.1016/s0015-0282(01)03275-7. PMID 11849631
- [Result] Zacur HA, Hedon B, Mansour D, Shangold GA, Fisher AC, Creasy GW. Integrated summary of Ortho Evra/Evra contraceptive patch adhesion in varied climates and conditions. Fertil Steril. 2002 Feb;77(2 Suppl 2):S32-5. doi: 10.1016/s0015-0282(01)03262-9. PMID 11849634